CLINICAL TRIAL: NCT00532272
Title: A Phase II Non-randomized, Parallel Group Study of Goserelin or Leuprorelin Plus Letrozole in Premenopausal Patients Versus Letrozole Alone in Postmenopausal Patients With Metastatic Breast Cancer
Brief Title: Goserelin/Letrozole in Premenopausal Patients vs Letrozole Alone in Postmenopausal Patients With MBC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: CENTER FOR BREAST CANCER, NATIONAL CANCER CENTER
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCCCTS-05-149
Record Dates: First submitted 2007-09-19; First posted 2007-09-20 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2007-09

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole; Goserelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- letrozole (Experimental): letrozole(2.5mg orally daily)
  Interventions: Drug: Letrozole ,Goserelin
- goserelin plus letrozole (Active Comparator): goserelin (3.6mg subcutaneously every 28 days) plus letrozole(2.5mg orally daily)
  Interventions: Drug: Letrozole ,Goserelin

INTERVENTIONS:
Drug: Letrozole ,Goserelin — Letrozole 2.5mg qd. Goserlin 3.6mg monthly(premenopausal)
  Other Names: Femara; Zoladex

SUMMARY:
Primary objective is to evaluate the response rates and clinical benefits of letrozole + goserelin in premenopausal patients versus letrozole alone in postmenopausal patients with metastatic breast cancer as first line hormonal therapy

DETAILED DESCRIPTION:
The sites of estrogen synthesis are the ovaries of premenopausal women and extragonadal sites such as fat, muscle, and skin, normal breast stromal cell and breast tumor tissue. After ovarian failure, estrogen is synthesized in peripheral tissues such as fat and muscles and this peripheral aromatization in postmenopausal women is almost completely inhibited by single-agent administration of the third generation inhibitor (anastrozole, letrozole and exemestane etc). In contrast, there is a barrier to using aromatase inhibitors as monotherapy in premenopausal women. First, high level of androstenedione competes initially with the inhibitors as substrate for the enzyme complex. Second, suppression of estrogen results in a reflex increase in gonadotrophin levels, provoking an ovarian hyperstimulation syndrome, which causes a steep increase of aromatase in the ovary and in turn overcomes the blockade by inhibitor.

The rationale of combination therapy regimen of a gonadotropins-releasing hormone (GnRH) agonist such as goserelin plus aromatase inhibitor in premenopausal patient is that, having effectively rendered the patients postmenopausal with the use of goserelin, the peripheral E2 production can be inhibited by aromatase inhibitor. Goserelin alone has been shown to produce castrate level of estradiol (E2) and response rates similar to oophorectomy in premenopausal women.

Selective aromatase inhibitors including letrozole have now become the standard second-line endocrine therapy, after the failure of tamoxifen in postmenopausal women with advanced breast cancer. Aromatase inhibitor is now challenged as first-line endocrine therapy for hormone-sensitive breast cancer.

Ovarian expression of aromatase is regulated by gonadotropins, LH and FSH. Theoretically, the combination of a GnRH analogue and an aromatase inhibitor can induce a complete estrogen blockade in premenopausal breast cancer patients. Although combination of goserelin and tamoxifen is an established therapeutic option in premenopausal patients with breast cancer, from the results of earlier studies comparing tamoxifen and aromatase inhibitors as first line therapy in postmenopausal patients with advanced breast cancer, it can be hypothesized that letrozole may accomplish better clinical results than tamoxifen as a first line hormonal therapy in patients with metastatic breast cancer who become menopause by GnRH agonist as first line hormonal therapy.

Developing this combination therapy would be particularly useful since more than 50% of breast cancers are developed in less than 50 years old women in Korea. Therefore, we are going to evaluate the clinical and endocrine results of first-line goserelin plus letrozole in premenopausal patients with metastatic breast cancer with first-line letrozole alone in postmenopausal patients.

Recently, CYP19 single nucleotide polymorphism (SNP) in tumor tissue was shown to be associated with the efficacy of aromatase inhibitor. In a study, when 67 postmenopausal patients with hormone receptor positive metastatic breast cancer were treated with letrozole, median TTP was significantly longer in patients with the rs4646 variant of intratumoral CYP19, a SNP in 3'-UTR, compared with normal CYP19 (17.2 months versus 6.4 months; P=0.02). This result suggests the importance of both the local aromatase activity and the tumor specific genetic alterations in the efficacy of aromatase inhibitors.

Up to recently, tumor-specific genetic markers have been assessed primarily in tumor biopsies. However, in advanced stage patients, tumor tissues are often unavailable, since surgery is not always performed or in some cases even the biopsy samples cannot be obtained, which limits the use of tumor tissue for genetic assessment. The detection of tumor specific genetic alterations in cancer patients at distant sites from the tumor, such as in blood, would provide a useful predictor for the efficacy to treatment. Some of the tumor genetic alterations have been observed in extracellular circulating DNA in blood samples of breast cancer patients, including alterations in microsatellites, LOH, TP53 gene mutations and so on.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically diagnosed stage IV or recurrent breast cancer patients according to American Joint Committee on Cancer (AJCC)
2. Positive estrogen receptor or progesterone receptor (>grade 3/7 by modified Allred IHC score)
3. Females at least 18 years of age and under 75 years
4. Prior chemotherapy for adjuvant setting or metastatic disease is allowed if the number of chemotherapy is ≤ 3.
5. Prior adjuvant antiestrogen therapy is allowed, provided that had not been received within 3 weeks before the entry of the study
6. Prior adjuvant aromatase inhibitor therapy is allowed if the agent had not been given within one year of the entry.
7. Prior radiation therapy is allowed as long as the irradiated area is not the only source of measurable disease.
8. No other forms of cancer therapy, such as radiation, immunotherapy for at least 3 weeks before the enrollment in the study.
9. Performance status of 0, 1 and 2 on the ECOG criteria.
10. Clinically measurable disease, defined as unidimensionally measurable lesions with clearly defined margins on x-ray, CT scan, MRI or physical examination. Lesions serving as measurable disease must be at least 1 cm by 1 cm, as defined by x-ray, CT scan, MRI, or physical examination.
11. Bone only or pleural fluid only disease is included as long as evaluation for clinical benefit is possible.
12. Estimated life expectancy of at least 12 weeks.
13. Compliant patient who can be followed-up adequately.
14. Adequate hematologic (WBC count 3,000/mm3, platelet count 100,000/mm3), hepatic (bilirubin level 1.8 mg/dL, AST, ALT 2.0xULN, albumin 2.5 g/dL), and renal (creatinine concentration 1.5 mg/dL) function.
15. Informed consent from patient or patient's relative.
16. Childbearing women should use non-hormonal contraceptive method.

Exclusion Criteria:

1. Previous chemotherapy more than 3 including adjuvant therapy.
2. Second primary malignancy (except in situ carcinoma of the cervix or adequately treated basal cell carcinoma of the skin or prior malignancy treated more than 5 years ago without recurrence).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2005-10; Primary Completion 2008-04 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the response rates and clinical benefits of letrozole + goserelin in premenopausal patients versus letrozole alone in postmenopausal patients with metastatic breast cancer as first line hormonal therapy | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Jungsil Ro, MD,PhD, Principal Investigator — National Cancer Center, Korea
Locations (1):
- National Cancer Center, Goyang, South Korea